CLINICAL TRIAL: NCT07285837
Title: Effect of an Intensive Rehabilitation Protocol Combining Constraint-Induced Movement Therapy and Bimanual Training on Upper Limb Use and Gross Motor Function in Children and Adolescents With Cerebral Palsy
Brief Title: Intensive Rehabilitation Program for Upper Limb in Children and Adolescents With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Habil'Hand+
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CP children and adolescents (Experimental): The program is tailored to the child's age and care setting. Children aged 3 to 8 years : 2 weeks program over 10 days with a total of 60 hours of CIMT+ BIT in a day-hospital setting.
  Adolescents aged 9 to 17 years in day-hospital care : 2 weeks program over 10 days with a total of 80 hours of CIMT+ BIT in a day-hospital setting.
  Adolescents aged 9 to 17 years in inpatient care : 2 weeks program over 10 days with a total of 80 hours of CIMT+ BIT in inpatient care.
  Interventions: Other: Intensive Rehabilitation

INTERVENTIONS:
Other: Intensive Rehabilitation — Children aged 3 to 8 years : 2 weeks program over 10 days including two individual sessions and three group sessions per participant per day combining CIMT and BIT.
  Adolescents aged 9 to 17 years in day-hospital care/ in inpatient care: 2 weeks program over 10 days including two individual sessions and three group sessions per participant per day combining CIMT and BIT.
  Daily routines, and activities involve functional and playful motor tasks of progressively increasing difficulty.

SUMMARY:
Cerebral palsy is the most common motor disability in children. Individuals with CP often experience significant difficulties in the use of their upper limbs, which affects their autonomy and quality of life. Conventional rehabilitation, although essential, is often insufficient to compensate for these deficits in a meaningful way.

The French National Authority for Health has issued recommendations for intensifying rehabilitation in order to maximize functional gains in children with CP. Among the intensive approaches that have been studied, two techniques have demonstrated efficacy: Constraint-Induced Movement Therapy (CIMT) and Bimanual Intensive Therapy (BIT).

CIMT focuses on restricting the use of the unaffected limb to encourage the use of the affected limb, thereby promoting neuroplasticity and functional improvement. In contrast, BIT emphasizes intensive training of both hands simultaneously to enhance coordination and overall upper limb functionality.

At the Ellen Poidatz Foundation, an intensive rehabilitation program has been developed that combines these two complementary approaches. This program, which is already in place, is based on the principles of neuromotor rehabilitation and motor learning. It integrates several methods recommended by the HAS, including Bimanual Intensive Therapy (BIT) such as HABIT (Grade A) or HABIT-ILE (Grade B), Modified Constraint-Induced Movement Therapy (mCIMT) (Grade B), and Adapted Physical Activity (APA) (Grade A).

The aim of this intensive program is to enhance the functional use of the upper limb by improving bimanual coordination, grasping, manipulation, and overall motor function. The program lasts 10 days over a 2-week period and is tailored to the child's age and care setting. It includes approximately 60 hours of rehabilitation for children aged 3 to 8 years and 80 hours for those aged 9 to 17 years, in line with current international recommendations.

The aim of this study is to evaluate the effectiveness of this existing intensive rehabilitation program in improving manual abilities in children with CP. Specifically, the study seeks to objectively assess the benefits of the Habil'Hand+ program and to contribute to the optimization of rehabilitation protocols for this population.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of CP mentioned in the medical record
* Aged between 3 and 17 years inclusive (<18 years)
* Global Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS) levels I to IV
* Ability to cooperate, understand and follow simple instructions
* Patient affiliated to the French social security system
* Voluntary patient whose parents have given their consent for their child to participate in the study.

Exclusion Criteria:

* Presence of injuries incompatible with participation in the program, or pain rated >3 on the Visual Analogue Scale (VAS)
* Presence of behavioral disorders
* History of botulinum toxin injections or surgical intervention within six months prior to study enrollment.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) /Both Hands Assessment(BoHA) | 3 months
  The AHA determine a score of natural use of the affected upper limb in standardized activity test. The BoHA is a standardized test designed for children with bilateral cerebral palsy. Both assessments contains 20 items rated on a 4-point scale (4=effective, 3=somewhat effective, 2=ineffective, and 1=does not do). A higher score therefore represents better performance.

SECONDARY OUTCOMES:
Melbourne Assessment 2 | 3 months
  Designed to evaluate four aspects of upper limb movement quality in children with neurological impairments: (1) range of motion, (2) accuracy of reach and placement, (3) dexterity in grasping, releasing, and manipulating objects, and (4) movement fluency. The full assessment includes 14 items, requiring the child to reach for, grasp, release, and manipulate simple objects.
Canadian Occupational Performance Measure (COPM) | 3 months
  Used to establish intervention goals that are consistent with the child's needs. The assessment is conducted in four steps: 1. Identification of occupational performance difficulties, 2. Prioritization of these difficulties according to their importance rated on a 10-point ordinal scale, 3. Rating of performance and satisfaction levels for the most important difficulties (up to five difficulties), using 10-point ordinal scales and 4. Re-evaluation (post-intervention) of performance and satisfaction levels for the difficulties identified at baseline.
Goal Attainment Scaling (GAS) | 3 months
  Used to evaluate the effectiveness of an intervention on individualized goals. The process involves the following steps: 1. Define specific goals - establish one or more precise, individualized objectives. 2. Weight the goals - rate each goal according to its importance and level of difficulty. 3.Define expected outcomes - specify the anticipated performance for each goal. 4.Establish the baseline - record the child's initial level of performance for each goal. 5. Calculate the GAS score - quantify goal attainment post-intervention using the standardized GAS formula.
Children's Hand Experience Questionnaire (CHEQ) | 3 months
  Used to assess the spontaneous use of the affected upper limb during bimanual activities of daily living. The Mini-CHEQ is designed for children aged 3 to 8 years and evaluates 21 activities, while the CHEQ 2.0 is intended for children aged 6 to 18 years and assesses 27 activities. The activities are presented in a random order. The questionnaire provides information on whether the activities are performed independently and whether one or both hands are used.
Box and Blocks test | 3 months
  Used to evaluate unilateral gross manual dexterity. Participant must transfer, one by one, with one hand, a maximum number of cubes from one side to the other of the box in 1 minute. A higher score represents better performance.
Gross Motor Function Measure (GMFM) | 3 months
  Used to assess gross motor function in children with cerebral palsy. The GMFM-66 evaluates five dimensions: lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping.
6 minutes walking test | 3 months
  To quantify changes in gait parameters (speed, cadence, step length). The patient is instructed to walk for 6 minutes in an unobstructed corridor. The distance walked is recorded for the calculation of walking speed. Fatigue is assessed with a Borg scale and heart rate is continuously recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Fondation Ellen Poidatz Habil'Hand+ — https://www.fondationpoidatz.com/arrow-cp/